CLINICAL TRIAL: NCT03582540
Title: Study Assessing the Interest of the Double-guidewire Technique for Catheterization of the Common Bile Duct.
Brief Title: Early Versus Delayed Double-guidewire Technique in Difficult Biliary Cannulation. (DFG)
Acronym: DFG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société Française d'Endoscopie Digestive (Other)
Responsible Party: Principal Investigator, Dr Arthur Laquiere, Gastroenterologist, Société Française d'Endoscopie Digestive
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ID RCB: 2016-A01016-45
Record Dates: First submitted 2018-06-28; First posted 2018-07-11 (Actual); Last update posted 2019-09-23 (Actual); Status verified 2018-06

CONDITIONS: Catheterization; Cholangiopancreatography; Endoscopic Retrograde Cholangiography; Biliary Cannulation; Difficult Biliary Cannulation; Double-guidewire Technique

STUDY DESIGN:
Intervention Model Description: Patients with a difficult biliary cannulation are included in the study if the guidewire is inserted in the pancreatic duct. At that point, patients are randomized in two arms: early versus delayed DGT. The early arm attempts biliary cannulation using the DGT immediately and the delayed arm uses the DGT only if 10 more minutes of conventional cannulation technique does not allow biliary cannulation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- early double-guidewire technique (DGT) (Active Comparator): First arm: early double-guidewire technique The early arm attempts biliary cannulation using the DGT immediately once the guidewire is inserted in the pancreatic duct in cases of difficult biliary cannulation.
  Interventions: Procedure: Double-guidewire cannulation technique
- delayed double-guidewire technique (DGT) (Active Comparator): In the delayed arm, once the guidewire is inserted in the pancreatic duct, the operator continues to attempt biliary cannulation with conventional technique (contrast- or guidewire-assisted). DGT is used only if 10 more minutes of conventional cannulation technique does not allow biliary access.
  Interventions: Procedure: Double-guidewire cannulation technique

INTERVENTIONS:
Procedure: Double-guidewire cannulation technique — With the DGT, a guidewire is first inserted deep into the PD. The cannulation device is then withdrawn, reloaded with a second guidewire, and reinserted through the working channel of the endoscope to cannulate the common bile duct.

SUMMARY:
This is a prospective randomized comparative multicentric study. Briefly, we will analyze the technical success, performance and clinical outcomes of early versus delayed double-guidewire technique (DGT) in difficult biliary cannulation.

DETAILED DESCRIPTION:
This is a prospective study performed in 20 tertiary medical centers in France. We aim to recruit 150 patients from 2016 to 2020. Patients with a native papilla scheduled for ERCP (endoscopic retrograde cholangiopancreatography) are screened for the study. Patients with a difficult biliary cannulation are included in the study if the guidewire is inserted in the pancreatic duct. At that point, patients are randomized in two arms: early versus delayed DGT. The early arm attempts biliary cannulation using the double-guidewire technique immediately and the delayed arm uses the double-guidewire technique only if 10 more minutes of standard cannulation technique does not allow biliary cannulation. The primary outcome is the biliary cannulation rate success. Secondary outcomes are complications rate and performance of the technique in both arms. Follow-up is 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years old and more
* Native papilla
* Clinical indications of ERCP
* Difficult biliary cannulation defined by unintentional guidewire insertion into the pancreatic duct before biliary cannulation is successful
* Informed consent completed by the patient

Exclusion Criteria:

* Contraindication to upper gastrointestinal endoscopy
* ERCP with direct biliary cannulation success
* ERCP with inability to cannulate the bile duct nor the pancreatic duct
* Coagulation or hemostasis disorder (TP < 60%, TCA> 40 sec. et plaquettes < 60000/mm3).
* Patient under active antiaggregant or anticoagulant medication other than aspirin
* Endoscopic treatment of chronic pancreatitis
* Pregnancy or breastfeeding
* ERCP performed by another operator than an investigator
* Patient's voluntary withdrawal
* Withdrawal decision by the investigator or sponsor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2016-11-02 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Biliary cannulation success rate | During the ERCP procedure
  The percentage of biliary cannulation success in both arms.

SECONDARY OUTCOMES:
Immediate morbidity | From the start, until 30 minutes after completion of ERCP
  Any complications (procedure related, clinical or anesthesiological) occurring during the procedure or during the immediate post-intervention period.
Delayed morbidity | 30 minutes after ERCP completion and up to 30 days
  Morbidities occurring more than 30 minutes and up to 1 month after ERCP completion. Special attention will be taken for bowel perforation, gastrointestinal bleeding and acute pancreatitis
procedural time | time from the first guidewire insertion into the pancreatic duct up to the end of cannulation.
  The time taken in minutes between patient randomization (at the first guidewire insertion into the pancreatic duct) and successful biliary cannulation.

CONTACTS AND LOCATIONS:
Overall Officials: ARTHUR LAQUIERE, MD, Principal Investigator — Société Française d'Endoscopie Digestive
Locations (8):
- France (8):
  - Clinique de Bercy, Charenton-le-Pont
  - Hôpital Dupuytren, Limoges
  - Hopital Saint Joseph, Marseille
  - Groupe Hospitalier Diaconesses - La Croix Saint-Simon, Paris
  - Hôpital Haut Lévêque, Pessac
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Centre Hospitalier de Bigorre, Tarbes
  - Centre Hospitalier de Vichy, Vichy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Adler DG, Baron TH, Davila RE, Egan J, Hirota WK, Leighton JA, Qureshi W, Rajan E, Zuckerman MJ, Fanelli R, Wheeler-Harbaugh J, Faigel DO; Standards of Practice Committee of American Society for Gastrointestinal Endoscopy. ASGE guideline: the role of ERCP in diseases of the biliary tract and the pancreas. Gastrointest Endosc. 2005 Jul;62(1):1-8. doi: 10.1016/j.gie.2005.04.015. No abstract available. PMID 15990812
- [Result] Freeman ML, Guda NM. ERCP cannulation: a review of reported techniques. Gastrointest Endosc. 2005 Jan;61(1):112-25. doi: 10.1016/s0016-5107(04)02463-0. No abstract available. PMID 15672074
- [Result] Hisa T, Matsumoto R, Takamatsu M, Furutake M. Impact of changing our cannulation method on the incidence of post-endoscopic retrograde cholangiopancreatography pancreatitis after pancreatic guidewire placement. World J Gastroenterol. 2011 Dec 28;17(48):5289-94. doi: 10.3748/wjg.v17.i48.5289. PMID 22219598
- [Result] Freeman ML, DiSario JA, Nelson DB, Fennerty MB, Lee JG, Bjorkman DJ, Overby CS, Aas J, Ryan ME, Bochna GS, Shaw MJ, Snady HW, Erickson RV, Moore JP, Roel JP. Risk factors for post-ERCP pancreatitis: a prospective, multicenter study. Gastrointest Endosc. 2001 Oct;54(4):425-34. doi: 10.1067/mge.2001.117550. PMID 11577302
- [Result] Artifon EL, Sakai P, Cunha JE, Halwan B, Ishioka S, Kumar A. Guidewire cannulation reduces risk of post-ERCP pancreatitis and facilitates bile duct cannulation. Am J Gastroenterol. 2007 Oct;102(10):2147-53. doi: 10.1111/j.1572-0241.2007.01378.x. Epub 2007 Jun 20. PMID 17581267
- [Result] Cennamo V, Fuccio L, Repici A, Fabbri C, Grilli D, Conio M, D'Imperio N, Bazzoli F. Timing of precut procedure does not influence success rate and complications of ERCP procedure: a prospective randomized comparative study. Gastrointest Endosc. 2009 Mar;69(3 Pt 1):473-9. doi: 10.1016/j.gie.2008.09.037. PMID 19231488
- [Result] Cennamo V, Fuccio L, Zagari RM, Eusebi LH, Ceroni L, Laterza L, Fabbri C, Bazzoli F. Can early precut implementation reduce endoscopic retrograde cholangiopancreatography-related complication risk? Meta-analysis of randomized controlled trials. Endoscopy. 2010 May;42(5):381-8. doi: 10.1055/s-0029-1243992. Epub 2010 Mar 19. PMID 20306386
- [Result] Parlak E, Cicek B, Disibeyaz S, Kuran S, Sahin B. Early decision for precut sphincterotomy: is it a risky preference? Dig Dis Sci. 2007 Mar;52(3):845-51. doi: 10.1007/s10620-006-9546-x. PMID 17273923
- [Result] Slivka A. A new technique to assist in bile duct cannulation. Gastrointest Endosc. 1996 Nov;44(5):636. doi: 10.1016/s0016-5107(96)70038-x. No abstract available. PMID 8934189
- [Result] Gotoh Y, Tamada K, Tomiyama T, Wada S, Ohashi A, Satoh Y, Higashizawa T, Miyata T, Ido K, Sugano K. A new method for deep cannulation of the bile duct by straightening the pancreatic duct. Gastrointest Endosc. 2001 Jun;53(7):820-2. doi: 10.1067/mge.2001.113387. No abstract available. PMID 11375604
- [Result] Vandervoort J, Soetikno RM, Tham TC, Wong RC, Ferrari AP Jr, Montes H, Roston AD, Slivka A, Lichtenstein DR, Ruymann FW, Van Dam J, Hughes M, Carr-Locke DL. Risk factors for complications after performance of ERCP. Gastrointest Endosc. 2002 Nov;56(5):652-6. doi: 10.1067/mge.2002.129086. PMID 12397271
- [Result] Caletti GC, Vandelli A, Bolondi L, Fontana G, Labo G. Endoscopic retrograde cholangiography (ERC) through artificial endoscopic choledocho-duodenal fistula. Endoscopy. 1978 Aug;10(3):203-6. doi: 10.1055/s-0028-1098295. PMID 699889
- [Result] Siegel JH. Precut papillotomy: a method to improve success of ERCP and papillotomy. Endoscopy. 1980 May;12(3):130-3. doi: 10.1055/s-2007-1021728. PMID 7379762
- [Result] Osnes M, Kahrs T. Endoscopic choledochoduodenostomy for choledocholithiasis through choledochoduodenal fistula. Endoscopy. 1977 Aug;9(3):162-5. doi: 10.1055/s-0028-1098510. PMID 913369
- [Result] Dumonceau JM, Deviere J, Cremer M. A new method of achieving deep cannulation of the common bile duct during endoscopic retrograde cholangiopancreatography. Endoscopy. 1998 Sep;30(7):S80. doi: 10.1055/s-2007-1001379. No abstract available. PMID 9826155
- [Result] Angsuwatcharakon P, Rerknimitr R, Ridtitid W, Ponauthai Y, Kullavanijaya P. Success rate and cannulation time between precut sphincterotomy and double-guidewire technique in truly difficult biliary cannulation. J Gastroenterol Hepatol. 2012 Feb;27(2):356-61. doi: 10.1111/j.1440-1746.2011.06927.x. PMID 21916994
- [Result] Cote GA, Mullady DK, Jonnalagadda SS, Keswani RN, Wani SB, Hovis CE, Ammar T, Al-Lehibi A, Edmundowicz SA, Komanduri S, Azar RR. Use of a pancreatic duct stent or guidewire facilitates bile duct access with low rates of precut sphincterotomy: a randomized clinical trial. Dig Dis Sci. 2012 Dec;57(12):3271-8. doi: 10.1007/s10620-012-2269-2. Epub 2012 Jun 26. PMID 22732831
- [Result] Herreros de Tejada A, Calleja JL, Diaz G, Pertejo V, Espinel J, Cacho G, Jimenez J, Millan I, Garcia F, Abreu L; UDOGUIA-04 Group. Double-guidewire technique for difficult bile duct cannulation: a multicenter randomized, controlled trial. Gastrointest Endosc. 2009 Oct;70(4):700-9. doi: 10.1016/j.gie.2009.03.031. Epub 2009 Jun 27. PMID 19560764
- [Result] Yoo YW, Cha SW, Lee WC, Kim SH, Kim A, Cho YD. Double guidewire technique vs transpancreatic precut sphincterotomy in difficult biliary cannulation. World J Gastroenterol. 2013 Jan 7;19(1):108-14. doi: 10.3748/wjg.v19.i1.108. PMID 23326171
- [Result] Xinopoulos D, Bassioukas SP, Kypreos D, Korkolis D, Scorilas A, Mavridis K, Dimitroulopoulos D, Paraskevas E. Pancreatic duct guidewire placement for biliary cannulation in a single-session therapeutic ERCP. World J Gastroenterol. 2011 Apr 21;17(15):1989-95. doi: 10.3748/wjg.v17.i15.1989. PMID 21528077
- [Result] Lee TH, Hwang SO, Choi HJ, Jung Y, Cha SW, Chung IK, Moon JH, Cho YD, Park SH, Kim SJ. Sequential algorithm analysis to facilitate selective biliary access for difficult biliary cannulation in ERCP: a prospective clinical study. BMC Gastroenterol. 2014 Feb 17;14:30. doi: 10.1186/1471-230X-14-30. PMID 24529239
- [Result] Goff JS. Long-term experience with the transpancreatic sphincter pre-cut approach to biliary sphincterotomy. Gastrointest Endosc. 1999 Nov;50(5):642-5. doi: 10.1016/s0016-5107(99)80012-1. PMID 10536319
- [Result] Tang SJ, Haber GB, Kortan P, Zanati S, Cirocco M, Ennis M, Elfant A, Scheider D, Ter H, Dorais J. Precut papillotomy versus persistence in difficult biliary cannulation: a prospective randomized trial. Endoscopy. 2005 Jan;37(1):58-65. doi: 10.1055/s-2004-826077. PMID 15657860
- [Derived] Laquiere A, Privat J, Jacques J, Legros R, Urena-Campos R, Belkhodja H, Subtil C, Kanafi L, Lecomte L, Boustiere C, Katsogiannou M, Karsenti D. Early double-guidewire versus repeated single-guidewire technique to facilitate selective bile duct cannulation: a randomized controlled trial. Endoscopy. 2022 Feb;54(2):120-127. doi: 10.1055/a-1395-7485. Epub 2021 Apr 15. PMID 33860484